CLINICAL TRIAL: NCT05330871
Title: A Single Center, Open-label, Parallel Controlled, Randomized Phase II Study to Evaluate the Safety and Immunogenicity of Ad5-nCoV-IM, Ad5-nCoV-IH or Inactivated COVID-19 Vaccine in Population 6 to 17 Years of Age
Brief Title: Evaluate the Safety and Immunogenicity of Ad5 COVID-19 Vaccines for Booster Use in Children Aged 6-17 Years.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seventh Medical Center of PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-Ad5-nCoV-IH-#
Record Dates: First submitted 2022-04-14; First posted 2022-04-15 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Ad5; Heterologous; Safety; Immunogenicity; 6-17 years; Inactivated COVID-19 vaccine; boost
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5 | interventions — Inhalation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- 1. Adolescent booster sentinel group (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 1 Nebulized inhalation for booster groups
- 2. Adolescent booster safety group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 2 Nebulized inhalation for booster groups
- 3. Adolescent booster immuno-persistency group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 3 Nebulized inhalation for booster groups
- 4. Adolescent booster cellular immunity group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 4 Nebulized inhalation for booster groups
- 5. Adolescent booster safety group to receive Ad5-nCoV-IM (Experimental): 1 dose of 0.3ml Ad5-nCoV-IM
  Interventions: Biological: 5 Intramuscular injection for booster groups
- 6. Adolescent booster immuno-persistency group to receive Ad5-nCoV-IM (Experimental): 1 dose of 0.3ml Ad5-nCoV-IM
  Interventions: Biological: 6 Intramuscular injection for booster groups
- 7. Adolescent booster cellular immunity group to receive Ad5-nCoV-IM (Experimental): 1 dose of 0.3ml Ad5-nCoV-IM
  Interventions: Biological: 7 Intramuscular injection for booster groups
- 8. Adolesent booster safety group to receive ICV (Active Comparator): 1 dose of 0.5ml ICV
  Interventions: Biological: 8 Intramuscular injection for booster groups
- 9. Adolescent booster immunopersistency group to receive ICV (Active Comparator): 1 dose of 0.5ml ICV
  Interventions: Biological: 9 Intramuscular injection for booster groups
- 10. Adolescent booster cellular immunity group to receive ICV (Active Comparator): 1 dose of 0.5ml ICV
  Interventions: Biological: 10 Intramuscular injection for booster groups
- 11. Children booster sentinel group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 11 Nebulized inhalation for booster groups
- 12. Children booster safety group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 12 Nebulized inhalation for booster groups
- 13. Children booster immuno-persistency group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 13 Nebulized inhalation for booster groups
- 14. Children booster cellular immunity group to receive Ad5-nCoV-IH (Experimental): 1 dose of 0.1ml Ad5-nCoV-IH
  Interventions: Biological: 14 Nebulized inhalation for booster groups
- 15. Children booster safety group to receive Ad5-nCoV-IM (Experimental): 1 dose of 0.3ml Ad5-nCoV-IM
  Interventions: Biological: 15 Intramuscular injection for booster groups
- 16. Children booster immuno-persistency group to receive Ad5-nCoV-IM (Experimental): 1 dose of 0.3ml Ad5-nCoV-IM
  Interventions: Biological: 16 Intramuscular injection for booster groups
- 17. Children booster cellular immunity group to receive Ad5-nCoV-IM (Experimental): 1 dose of 0.3ml Ad5-nCoV-IM
  Interventions: Biological: 17 Intramuscular injection for booster groups
- 18. Children booster safety group to receive ICV (Active Comparator): 1 dose of 0.5ml ICV
  Interventions: Biological: 18 Intramuscular injection for booster groups
- 19. Children booster immuno-persistency group to receive ICV (Active Comparator): 1 dose of 0.5ml ICV
  Interventions: Biological: 19 Intramuscular injection for booster groups
- 20. Children booster cellular immunity group to receive ICV (Active Comparator): 1 dose of 0.5ml ICV
  Interventions: Biological: 20 Intramuscular injection for booster groups
- 21. Adolescent primary sentinel group (Experimental): 2 doses of 0.1ml Ad5-nCoV-IH, 56 days interval
  Interventions: Biological: 21 Nebulized inhalation for primary groups
- 22. Adolescent primary group (Experimental): 2 doses of 0.1ml Ad5-nCoV-IH, 56 days interval
  Interventions: Biological: 22 Nebulized inhalation for primary groups
- 23. Children primary sentinel group (Experimental): 2 doses of 0.1ml Ad5-nCoV-IH, 56 days interval
  Interventions: Biological: 23 Nebulized inhalation for primary groups
- 24. Children primary group (Experimental): 2 doses of 0.1ml Ad5-nCoV-IH, 56 days interval
  Interventions: Biological: 24 Nebulized inhalation for primary groups

INTERVENTIONS:
Biological: 1 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 1. Adolescent booster sentinel group
Biological: 2 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 2. Adolescent booster safety group to receive Ad5-nCoV-IH
Biological: 3 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 3. Adolescent booster immuno-persistency group to receive Ad5-nCoV-IH
Biological: 4 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 4. Adolescent booster cellular immunity group to receive Ad5-nCoV-IH
Biological: 5 Intramuscular injection for booster groups — Ad5-nCoV-IM, 1 dose 0.3ml
  Other Names: Recombinant Corona Virus Vaccine (Adenovirus Type 5 Vector)
  Arms: 5. Adolescent booster safety group to receive Ad5-nCoV-IM
Biological: 6 Intramuscular injection for booster groups — Ad5-nCoV-IM, 1 dose 0.3ml
  Other Names: Recombinant Corona Virus Vaccine (Adenovirus Type 5 Vector)
  Arms: 6. Adolescent booster immuno-persistency group to receive Ad5-nCoV-IM
Biological: 7 Intramuscular injection for booster groups — Ad5-nCoV-IM, 1 dose 0.3ml
  Other Names: Recombinant Corona Virus Vaccine (Adenovirus Type 5 Vector)
  Arms: 7. Adolescent booster cellular immunity group to receive Ad5-nCoV-IM
Biological: 8 Intramuscular injection for booster groups — ICV, 1 dose 0.5ml
  Other Names: Inactivated COVID-19 Vaccine
  Arms: 8. Adolesent booster safety group to receive ICV
Biological: 9 Intramuscular injection for booster groups — ICV, 1 dose 0.5ml
  Other Names: Inactivated COVID-19 Vaccine
  Arms: 9. Adolescent booster immunopersistency group to receive ICV
Biological: 10 Intramuscular injection for booster groups — 1 dose 0.5ml
  Other Names: Inactivated COVID-19 Vaccine
  Arms: 10. Adolescent booster cellular immunity group to receive ICV
Biological: 11 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 11. Children booster sentinel group to receive Ad5-nCoV-IH
Biological: 12 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 12. Children booster safety group to receive Ad5-nCoV-IH
Biological: 13 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 13. Children booster immuno-persistency group to receive Ad5-nCoV-IH
Biological: 14 Nebulized inhalation for booster groups — Ad5-nCoV-IH, 1 dose 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 14. Children booster cellular immunity group to receive Ad5-nCoV-IH
Biological: 15 Intramuscular injection for booster groups — Ad5-nCoV-IM, 1 dose 0.3ml
  Other Names: Recombinant Corona Virus Vaccine (Adenovirus Type 5 Vector)
  Arms: 15. Children booster safety group to receive Ad5-nCoV-IM
Biological: 16 Intramuscular injection for booster groups — Ad5-nCoV-IM, 1 dose 0.3ml
  Other Names: Recombinant Corona Virus Vaccine (Adenovirus Type 5 Vector)
  Arms: 16. Children booster immuno-persistency group to receive Ad5-nCoV-IM
Biological: 17 Intramuscular injection for booster groups — Ad5-nCoV-IM, 1 dose 0.3ml
  Other Names: Recombinant Corona Virus Vaccine (Adenovirus Type 5 Vector)
  Arms: 17. Children booster cellular immunity group to receive Ad5-nCoV-IM
Biological: 18 Intramuscular injection for booster groups — ICV, 1 dose 0.5ml
  Other Names: Inactivated COVID-19 Vaccine
  Arms: 18. Children booster safety group to receive ICV
Biological: 19 Intramuscular injection for booster groups — ICV, 1 dose 0.5ml
  Other Names: Inactivated COVID-19 Vaccine
  Arms: 19. Children booster immuno-persistency group to receive ICV
Biological: 20 Intramuscular injection for booster groups — ICV, 1 dose 0.5ml
  Other Names: Inactivated COVID-19 Vaccine
  Arms: 20. Children booster cellular immunity group to receive ICV
Biological: 21 Nebulized inhalation for primary groups — Ad5-nCoV-IH, 2 doses 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 21. Adolescent primary sentinel group
Biological: 22 Nebulized inhalation for primary groups — Ad5-nCoV-IH, 2 doses 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 22. Adolescent primary group
Biological: 23 Nebulized inhalation for primary groups — Ad5-nCoV-IH, 2 doses 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 23. Children primary sentinel group
Biological: 24 Nebulized inhalation for primary groups — Ad5-nCoV-IH, 2 doses 0.1ml
  Other Names: Recombinant COVID-19 Vaccine for Inhalation
  Arms: 24. Children primary group

SUMMARY:
This is a single center, open-label, parallel controlled, and randomized Phase II clinical trial to evaluate the safety and immunogenicity of two types of Recombinant Novel Corona Virus Vaccine (Adenovirus type 5 vector) in population aged 6-17 years who have been previously immunized with 2 doses of inactivated COVID-19 vaccine. This is to evaluate the safety and immunogenicity of different heterologous prime-boost regimen in this population.

DETAILED DESCRIPTION:
Participants will be randomized into two age groups: children aged 6-12 years and adolescents aged 13-17 years. Subjects who have previously been immunized with 2 doses of inactivated COVID-19 vaccine will be randomized into the booster dose groups to receive either 1 dose of 0.1ml inhaled Ad5- nCoV-IH, 1 dose of 0.3ml intramuscular Ad5-nCoV-IM or 1 dose of 0.5ml intramuscular inactivated vaccine ICV as activecomparator in a ratio of 3:1:1. Participants who have not received any COVID-19 vaccine previously will be randomized into 2 primary dose age groups: children aged 6-12 years and adolescents aged 13-17 years to receive 2 doses of 0.1ml inhaled Ad5-nCoVIH. The first 5 subjects of each age group will enter the sentinel group to receive Ad5-nCoV-IH and monitor for safety before the rest of the enrollment process.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 6-17 years at the time of enrollment.
* Obtain written informed assent from participants and consent from parents, guardians or legal representatives.
* Able and willing to complete all the scheduled study procedures during the whole study follow-up period of 12 months.
* Have not received any COVID-19 vaccines (for primary groups only).

Exclusion Criteria:

* Medical or family history of seizures, epilepsy, encephalopathy, and psychosis disorders.
* History of allergies to any ingredient of Ad5-nCoV, history of serious allergic reactions to any vaccine, history of allergies and asthma.
* History of vaccine related SAEs after receiving any COVID-19 vaccines.
* Positive urine pregnancy test result, females with child bearing potential (have had menarche).
* Acute febrile diseases and infectious diseases, medical history of SARS (SARS-CoV-1).
* Axillary temperature >37.0#.
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and uncontrollable by medications.
* Severe chronic diseases or with advanced stage conditions which cannot be controlled smoothly, such as diabetes, thyroid disease, etc.
* Congenital or acquired angioedema/neurological edema.
* Urticaria history within 1 year before receiving the study vaccine.
* Asplenia or functional aspleenia.
* Thrombocytopenia or other coagulation disorders (may cause contraindications for intramuscular injection).
* Trypanophobia.
* Severe nasal or oral diseases, such as acute rhinitis (sinusitis), allergic rhinitis, oral ulcers, throat redness, and swelling.
* Lung function abnormalities such as chronic obstructive pulmonary disease and pulmonary fibrosis.
* Abnormal laboratory test indexes that are clinical significant as judged by the investigator (including white blood cell count, lymphocyte count, eosinophils, neutrophils, platelets, hemoglobin, alanine aminotransferase ALT, aspartate aminotransferase AST, total bilirubin , creatinine, activated partial thromboplastin time) (for sentinel and safety groups only).
* Respiratory rate ≥ 17 times per minute (for sentinel and safety groups only).
* History of receiving immunosuppressant therapy, anti-allergic therapy, cytotoxic therapy, nebulized corticosteroid therapy in the past 6 months (not including corticosteroid spray treatment for allergic rhinitis, and surface corticosteroid treatment for acute non-complicated dermatitis).
* Prior administration of blood products in last 4 months.
* Received other investigational drugs within 1 month before the study.
* Prior administration of live attenuated vaccines within 1 month before the study.
* Prior administration of subunit or inactivated vaccines within 14 days before the study.
* Current anti-tuberculosis therapy.
* Medical history of Covid-19 disease/infection.
* History of epidemiological exposure to COVID-19; have traveled to medium or high-risk areas in the past 21 days or have a history of travelling outside the country
* Any condition that in the opinion of the investigators may interfere with the participants' compliance or evaluation of study objectives or informed consent (i.e. medical, psychological, social or other conditions, etc).

Exclusion criteria for second dose:

* Newly emerged situations that meet the first-dose exclusion criteria.
* Vaccine related SAE post first dose vaccination.
* Serious allergic reactions post first dose vaccination.
* Other reasons in the opinion of the investigator.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 410 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of anti SARS-CoV-2 neutralizing antibody | 28 days post vaccination
  GMT of anti SARS-CoV-2 neutralizing antibody
Incidence of adverse reaction (AR) | 0-14 days post each vaccination
  Incidence of adverse reaction (AR)

SECONDARY OUTCOMES:
Immunogenicity of anti SARS-CoV-2 S protein IgG antibody | 28 days post vaccination
  Seroconversion rate of anti SARS-CoV-2 S protein IgG antibody (4 times fold increase)
Immunogenicity of anti SARS-CoV-2 S protein IgG antibody | 28 days post vaccination
  GMC of anti SARS-CoV-2 S protein IgG antibody
Immunogenicity of anti SARS-CoV-2 S protein IgG antibody | 28 days post vaccination
  GMI of anti SARS-CoV-2 S protein IgG antibody
Immunogenicity of anti Ad5 vector antibody | Day 0 before vaccination
  Stratified analysis of baseline level of anti Ad5 vector antibody
Immunogenicity of anti SARS-CoV-2 neutralizing antibody | Post vaccination
  Seroconversion rate of anti SARS-CoV-2 neutralizing antibody
Immunogenicity of anti SARS-CoV-2 neutralizing antibody | Post vaccination
  GMI of anti SARS-CoV-2 neutralizing antibody
Incidence of adverse event/adverse reaction | 30 minutes post each vaccination
  Incidence of AE/AR
Incidence of adverse event/adverse reaction | 0-28 days post each vaccination
  Incidence of AE/AR
Incidence of Serious Adverse Event | First dose vaccination to 12 months post last vaccination]
  Incidence of SAE
Changes in laboratory indicators in sentinel groups and safety groups | 4 days post each vaccination
  Changes in WBC counts
Changes in laboratory indicators in sentinel groups and safety groups | 4 days post each vaccination
  Changes in lymphocytes counts
Changes in laboratory indicators in sentinel groups and safety groups | 4 days post each vaccination
  Changes in platelet counts
Immuno-persistency of anti SARS-CoV-2 S protein IgG antibody | 3 months, 6 months and 12 months post vaccination
  GMC of anti SARS-CoV-2 S protein IgG antibody in immuno-persistency and primary groups
Immuno-persistency of anti SARS-CoV-2 S protein IgG antibody | 6 months and 12 months post vaccination
  Seroconversion rate of anti SARS-CoV-2 S protein IgG antibody in immuno-persistency and primary groups
Immuno-persistency of anti SARS-CoV-2 S protein IgG antibody | 6 months and 12 months post vaccination
  GMI of anti SARS-CoV-2 S protein IgG antibody in immuno-persistency and primary groups

CONTACTS AND LOCATIONS:
Overall Officials: Chen Dong, Study Chair — Seventh Medical Center of PLA General Hospital
Locations (1):
- CDC of of Luxi County, Xiangxi Tujia and Miao Autonomous Prefecture, Hunan Province, Xiangxi, Hunan, China

REFERENCES:
- [Derived] Huang T, Zhang S, Dai DF, Wang BS, Zhuang L, Huang HT, Wang ZF, Zhao JS, Li QP, Wu SP, Wang X, Zhang WD, Zhao ZH, Li H, Zhang YP, Yang XL, Jiang XY, Gou JB, Hou LH, Gao LD, Feng ZC. Safety and immunogenicity of heterologous boosting with orally aerosolised or intramuscular Ad5-nCoV vaccine and homologous boosting with inactivated vaccines (BBIBP-CorV or CoronaVac) in children and adolescents: a randomised, open-label, parallel-controlled, non-inferiority, single-centre study. Lancet Respir Med. 2023 Aug;11(8):698-708. doi: 10.1016/S2213-2600(23)00129-7. Epub 2023 May 17. PMID 37209700